CLINICAL TRIAL: NCT00530595
Title: Effects of Angiotensin Receptor Antagonist on Prohibiting Cardiovascular Events on Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saitama Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-01
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-09

CONDITIONS: Cardiovascular Disease
Keywords: hemodialysis
MeSH Terms: conditions — Cardiovascular Diseases | interventions — candesartan; Valsartan; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: candesartan or valsartan or losartan

SUMMARY:
Cardiovascular disease is a leading cause of mortality in patients on hemodialysis therapy (HD), accounting for 30 to 50% of all death. Although angiotensin receptor blockers (ARBs) are effective for patients with diabetes and chronic kidney disease in reducing or preventing cardiovascular diseases, there has been no decisive study that demonstrated treatment with ARBs is effective in patients on HD.

ELIGIBILITY:
Inclusion Criteria:

* 30 to 80 years of age
* Receiving hemodialysis at least 12 months and less than 5 years
* Pre-dialysis systolic blood pressure was more than 160 mmHg, or more than 150 mmHg if the patients received antihypertensive agents.

Exclusion Criteria:

* Use of angiotensin receptor blocker or angiotensin converting enzyme inhibitor

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Hiromichi Suzuki, MD, PhD, Study Director — Department of Nephrology, Saitama Medical University

REFERENCES:
- [Derived] Suzuki H, Kanno Y, Sugahara S, Ikeda N, Shoda J, Takenaka T, Inoue T, Araki R. Effect of angiotensin receptor blockers on cardiovascular events in patients undergoing hemodialysis: an open-label randomized controlled trial. Am J Kidney Dis. 2008 Sep;52(3):501-6. doi: 10.1053/j.ajkd.2008.04.031. Epub 2008 Jul 24. PMID 18653268